CLINICAL TRIAL: NCT00477919
Title: E-MOSAIC: A Multicenter Randomized Controlled Phase III Study of Longitudinal Electronic Monitoring of Symptoms and Syndromes Associated With Advanced Cancer in Patients Receiving Anticancer Treatment in Palliative Intention
Brief Title: E-MOSAIC Electronic Tool to Monitor Symptoms
Status: Completed | Type: Observational
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: SAKK 95/06; EU-20711
Record Dates: First submitted 2007-05-23; First posted 2007-05-24 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Cancer
Keywords: stage IV melanoma; stage IV renal cell cancer; unresectable extrahepatic bile duct cancer; advanced malignant mesothelioma; stage IV prostate cancer; adult giant cell glioblastoma; adult gliosarcoma; extensive stage small cell lung cancer; stage IV non-small cell lung cancer; stage IV colon cancer; stage IV gastric cancer; stage IV esophageal cancer; stage IV bladder cancer; male breast cancer; stage IV breast cancer; stage IV ovarian epithelial cancer; stage IV ovarian germ cell tumor; ovarian sarcoma; ovarian stromal cancer; fatigue; anorexia; cachexia; pain; weight changes; depression; poor performance status; recurrent adult brain tumor; clear cell sarcoma of the kidney; advanced adult primary liver cancer; recurrent adult primary liver cancer; recurrent small cell lung cancer; recurrent bladder cancer; recurrent breast cancer; recurrent colon cancer; recurrent esophageal cancer; recurrent gastric cancer; recurrent melanoma; recurrent non-small cell lung cancer; recurrent ovarian epithelial cancer; recurrent ovarian germ cell tumor; stage IV pancreatic cancer; recurrent prostate cancer; recurrent renal cell cancer; recurrent pancreatic cancer; stage IV rectal cancer; recurrent rectal cancer; recurrent malignant mesothelioma; recurrent carcinoma of unknown primary; stage IV adult soft tissue sarcoma; recurrent adult soft tissue sarcoma; stage IV uterine sarcoma; recurrent uterine sarcoma; recurrent extrahepatic bile duct cancer; unresectable gallbladder cancer; recurrent gallbladder cancer; adult glioblastoma
MeSH Terms: conditions — Neoplasms; Melanoma; Carcinoma, Renal Cell; Prostatic Neoplasms; Glioblastoma; Gliosarcoma; Carcinoma, Non-Small-Cell Lung; Colonic Neoplasms; Stomach Neoplasms; Esophageal Neoplasms; Urinary Bladder Neoplasms; Breast Neoplasms, Male; Breast Neoplasms; Carcinoma, Ovarian Epithelial; Fatigue; Anorexia; Cachexia; Pain; Body Weight Changes; Depression; Brain Neoplasms; Carcinoma, Hepatocellular; Small Cell Lung Carcinoma; Pancreatic Neoplasms; Rectal Neoplasms; Mesothelioma, Malignant; Neoplasms, Unknown Primary; Sarcoma; Bile Duct Neoplasms; Gallbladder Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Weekly assessment by E-MOSAIC: Patients complete a weekly assessment comprising visual analogue scales (VAS) of pain, fatigue, drowsiness, nausea, anxiety, depression, shortness of breath, loss of appetite, and overall well-being; up to 3 optional symptoms selected by the patient; and an estimated nutritional intake using an electronic tool for monitoring symptoms and syndromes associated with advanced cancer (E-MOSAIC). Nurses record the patient's weight, KPS score, body mass index, and assessment of current medication for pain (i.e., morphine-equivalent daily dose), fatigue, and anorexia/cachexia syndromes weekly. A Longitudinal Monitoring Sheet (LoMoS) is printed (comprising VAS of pain, pain medication, fatigue, KPS, medication for fatigue [i.e., methylphenidate hydrochloride or epoetin alfa], anorexia, weight change, nutritional intake, medication, supplements, counseling for anorexia, VAS of individually selected symptoms) and stored.
- Palm-based monitoring tool: Patients complete a weekly symptom assessment and nutritional intake using a Palm-based monitoring tool. Nurses record weight and Karnofsky performance status (KPS) scores weekly. A proof of electronic transfer sheet is printed and stored.

SUMMARY:
RATIONALE: A hand held electronic tool used to monitor symptoms and assess quality of life may improve communication between patients and their doctors and improve the ability to plan treatment for patients with advanced cancer receiving palliative care. It is not yet known whether symptoms are better controlled with or without use of this electronic tool.

PURPOSE: This randomized phase III trial is studying an electronic tool to see how well it records cancer symptoms in patients with advanced cancer receiving palliative care.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the effect of an electronic tool for monitoring symptoms and syndromes associated with advanced cancer (E-MOSAIC) and a Longitudinal Monitoring Sheet (LoMoS) on global quality of life (G-QOL) of patients with advanced incurable cancer receiving palliative anticancer treatment.

Secondary

* Determine if this tool affects communication between these patients and their treating physicians.
* Determine if this tool affects the symptoms and syndromes reported by these patients.
* Determine if this tool impacts symptom management performance.

Tertiary

* Identify factors influencing changes in G-QOL.
* Determine how patients adapt to illness and burden of treatment.
* Describe patients' decision-making preference.

OUTLINE: This is a controlled, randomized, longitudinal, multicenter study. Physicians are stratified according to participating center. Physicians are randomized to 1 of 2 arms. All patients allocated to a physician undergo the same intervention.

* Arm I: Patients complete a weekly symptom assessment and nutritional intake using a Palm-based monitoring tool. Nurses record weight and Karnofsky performance status (KPS) scores weekly. A proof of electronic transfer sheet is printed and stored.
* Arm II: Patients complete a weekly assessment comprising visual analogue scales (VAS) of pain, fatigue, drowsiness, nausea, anxiety, depression, shortness of breath, loss of appetite, and overall well-being; up to 3 optional symptoms selected by the patient; and an estimated nutritional intake using an electronic tool for monitoring symptoms and syndromes associated with advanced cancer (E-MOSAIC). Nurses record the patient's weight, KPS score, body mass index, and assessment of current medication for pain (i.e., morphine-equivalent daily dose), fatigue, and anorexia/cachexia syndromes weekly. A Longitudinal Monitoring Sheet (LoMoS) is printed (comprising VAS of pain, pain medication, fatigue, KPS, medication for fatigue [i.e., methylphenidate hydrochloride or epoetin alfa], anorexia, weight change, nutritional intake, medication, supplements, counseling for anorexia, VAS of individually selected symptoms) and stored.

In both arms, patients are assessed for outcome criteria at baseline and at weeks 3 and 6 (end of study).

PROJECTED ACCRUAL: A total of 24 physicians and 192 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of advanced incurable cancer
* Symptomatic disease, defined as meeting ≥ 1 of the following criteria:

  * Pain Visual Analogue Scale (VAS) ≥ 3/10 and/or morphine equivalent daily dose of ≥ 10 mg for ≥ 3 days
  * Anorexia VAS ≥ 3/10 and/or weight loss of ≥ 2% in 2 months or ≥ 5% in 6 months
  * Fatigue VAS ≥ 3/10 and/or Karnofsky performance status < 70%
  * Depression or anxiety VAS ≥ 3/10 and/or treatment with antidepressants for ≥ 5 days and planned for ≥ 1 month
* Receiving continuously, weekly, or biweekly palliative anticancer treatment meeting 1 of the following criteria:

  * At least 1 first-line treatment for any of the following:

    * Metastatic melanoma
    * Renal cell cancer
    * Pancreatic cancer
    * Biliary tract cancer
    * Mesothelioma
    * Prostate cancer (chemotherapy)
    * Advanced glioblastoma
  * At least 1 second-line treatment for any of the following:

    * Extensive stage small cell lung cancer
    * Stage IV non-small cell lung cancer
    * Colorectal cancer
    * Gastric cancer
    * Esophageal cancer
    * Bladder cancer
    * Sarcoma
    * Carcinoma of unknown primary
  * At least 1 third-line chemotherapy regimen for any of the following:

    * Metastatic breast cancer
    * Ovarian cancer
* Anticancer treatment must be given in an outpatient setting, not within a clinical trial, with weekly monitoring, and expected tumor response rate ≤ 20% according to the literature
* No testicular cancer
* No hematological malignancies
* No primary brain tumors other than glioblastoma
* Physician characteristics:

  * No change to standard of care for symptom assessment or to major communication skills strategies within the past 3 months
  * Experienced in medical oncology (i.e., worked ≥ 50% in clinical oncology within the past 24 months)
  * Likely to stay in the participating institution for the time required to treat ≥ 5 study patients
  * Able to independently communicate with the patient about all aspects of cancer care
  * Able to independently perform immediate changes of interventions in patient care without the institutional requirement to counsel another colleague before prescribing (i.e., for symptom control)
  * Completed a basic communication skills course or equivalent training (i.e., familiar with communication skills)

PATIENT CHARACTERISTICS:

* Able to understand assessment instrument language
* Able to understand physician communication without difficulty (i.e., due to culture, language, speech)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No concurrent participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced incurable cancer
Sampling Method: Probability Sample
Enrollment: 264 (Actual)
Dates: Start 2007-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Determine the effect of an electronic tool for monitoring symptoms and syndromes associated with advanced cancer (E-MOSAIC) and a Longitudinal Monitoring Sheet (LoMoS) on global quality of life (G-QOL) | Until trial ends

SECONDARY OUTCOMES:
Determine if this tool affects communication between these patients and their treating physicians. | Until trial ends
Determine if this tool affects the symptoms and syndromes reported by these patients | Until trial ends
Determine if this tool impacts symptom management performance | Until trial ends

CONTACTS AND LOCATIONS:
Overall Officials: Florian Strasser, MD, ABHPM, Study Chair — Cantonal Hospital of St. Gallen
Locations (7):
- Switzerland (7):
  - Universitaetsspital-Basel, Basel
  - Istituto Oncologico della Svizzera Italiana - Ospedale San Giovanni, Bellinzona
  - Inselspital Bern, Bern
  - Spital Buelach, Bülach
  - Kantonsspital Graubuenden, Chur
  - Kantonsspital Freiburg, Fribourg
  - Kantonsspital - St. Gallen, Sankt Gallen

REFERENCES:
- [Result] Blum D, Koeberle D, Ribi K, Schmitz SF, Utiger U, Klingbiel D, Strasser F. Electronic monitoring of symptoms and syndromes associated with cancer: methods of a randomized controlled trial SAKK 95/06 E-MOSAIC. BMC Palliat Care. 2012 Sep 24;11:19. doi: 10.1186/1472-684X-11-19. PMID 23006802
- [Result] Strasser F, Blum D, von Moos R, Cathomas R, Ribi K, Aebi S, Betticher D, Hayoz S, Klingbiel D, Brauchli P, Haefner M, Mauri S, Kaasa S, Koeberle D; Swiss Group for Clinical Cancer Research (SAKK). The effect of real-time electronic monitoring of patient-reported symptoms and clinical syndromes in outpatient workflow of medical oncologists: E-MOSAIC, a multicenter cluster-randomized phase III study (SAKK 95/06). Ann Oncol. 2016 Feb;27(2):324-32. doi: 10.1093/annonc/mdv576. Epub 2015 Dec 8. PMID 26646758